CLINICAL TRIAL: NCT01336998
Title: Administration of Arginine Supplementation in Preterm Infants and Measurement of Fecal Calprotectin as an Inflammatory Marker of the Intestine
Brief Title: Administration of Arginine Supplementation in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandra Hospital, Athens, Greece (Other)
Collaborators: University of Athens (Other)
Responsible Party: Elena Polycarpou/ MD, Pediatrician, Alexandra Hospital Athens Greece
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALEXANDRA 9159
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Necrotizing Enterocolitis
Keywords: necrotizing enterocolitis; arginine supplementation; calprotectin
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: arginine — oral L-arginine supplementation 261mg/kg/day (1,5mmol/kg/day), one dose daily ,from the 3rd day of life until the 28th day of life
  Other Names: L-arginine Nutricia

SUMMARY:
Calprotectin is a cytosolic component of neutrophils .Fecal calprotectin(FC) is a useful marker for exacerbation of inflammatory bowel disease in children .FC may be a useful marker for necrotizing enterocolitis (NEC).

NEC is one of the most common ,deadliest and enigmatic intestinal problems encountered mostly in premature infants. The precise pathophysiology of NEC is unclear ,but major factors thought to play an important role include an immature intestine ,an inflammatory response to intestinal microbes,enteral feedings and intestinal ischemia-reperfusion injury.Diagnosis of NEC is not easy clinically and up to now there is not a simple laboratory test to differentiate NEC at an early stage from other conditions in the neonate.

Arginine is the substrate for NO production in the gut and its deficiency may cause vasoconstriction and gut injury and thus predispose to NEC. In previous studies arginine supplementation was found to reduce the incidence of NEC in premature infants but more studies are needed for the use of arginine supplementation for the prevention of NEC.

The investigators aim is to measure the fecal calprotectin in very low birth weight (VLBW) infants during the first month of life as an inflammatory marker of the bowel and evaluate whether premature infants receiving arginine supplements had lower calprotectin values compared to the premature infants that did not .

The investigators hypothesize that arginine supplementation in preterm infants reduces the inflammation of the gut which will be shown by the lower fecal calprotectin values of the premature infants receiving arginine supplementation.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates born at Alexandra hospital during the study period
* < 34 weeks gestational age
* < 1500gr birth weight

Exclusion Criteria:

* major congenital abnormalities
* inborn errors of metabolism
* parents not consent

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
fecal calprotectin levels | first 28 days of life

SECONDARY OUTCOMES:
necrotizing enterocolitis | first 3 months of life
  the incidence of necrotizing enterocolitis in the study group

CONTACTS AND LOCATIONS:
Overall Officials: Kostalos Chistos, MD Phd, Study Chair — Alexandra Hospital neonatal intensive care unit
Locations (1):
- Alexandra Hospital, Athens, Athens, Greece